CLINICAL TRIAL: NCT06640114
Title: A Randomised Pilot Study of the Efficacy and Safety of Using Hemoperfusion With Efferon CT to Treat Patients With Severe Psoriasis
Brief Title: Hemoperfusion With Efferon CT for the Treatment of Patients With Severe Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-ct-2024-02
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; Hemoperfusion; Extracorporeal therapy; Cytokine adsorption
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Allocation of patients into groups will be done by stratified 1:1 randomisation.
  Stratification will be done by the patient's PASI index score (10 to 19, and more than 19).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline therapy (No Intervention): Patients who received only standard therapy according to the underlying disease (topical therapy, systemic therapy, phototherapy).
- Baseline therapy + Efferon CT (Experimental): Patients with moderate to severe psoriasis who were receiving standard therapy for the treatment of the underlying disease and who also received a single course of haemoperfusion with Efferon CT
  Interventions: Device: Efferon CT

INTERVENTIONS:
Device: Efferon CT — Efferon CT (JSC Efferon, Moscow, RF) is a device for extracorporeal blood purification by direct hemoperfusion. Detoxification is carried out by sorption of cytokines and other products of endogenous intoxication with a molecular size of up to 55 kDa.
  The duration of hemoperfusion is from 2 to 6 hours through peripheral venous access, followed by follow-up for 4 hours. The rate of hemoperfusion is from 60 to 80 ml/min. Anticoagulation is systemic (heparin).
  Arms: Baseline therapy + Efferon CT

SUMMARY:
Psoriasis is a chronic, inflammatory skin condition driven by the immune system, marked by red, scaly plaques that commonly affect the scalp and nails. About 30% of psoriasis patients may develop psoriatic arthritis, especially those with severe psoriasis or lesions on the nails or scalp. Research has identified distinct cytokine gene expression patterns in skin versus synovial tissue, which may explain the differing responses to biologic therapies in these areas. Factors such as genetic predisposition, infections, obesity, and biomechanical stress can trigger disease onset, leading to the release of cytokines that activate both the innate and adaptive immune responses. This immune activation can cause synovitis, enthesitis, erosions, and lesions in both articular cartilage and skin.

Given the reviewed literature and evidence that hemoperfusion with Efferon CT can non-specifically adsorb excess cytokines and inflammatory mediators, our research team hypothesizes that cytokine sorption could have beneficial clinical effects for patients with severe and moderate psoriasis. This study aims to evaluate the efficacy and safety of anticytokine hemoperfusion using the Efferon CT device for treating these patients.

DETAILED DESCRIPTION:
Psoriasis is a chronic, inflammatory, immune-mediated skin disease characterised by the appearance of erythematous and scaly plaques, often involving the scalp and nails. Approximately 30% of patients with psoriasis may develop psoriatic arthritis, particularly in patients with severe psoriasis or lesions on the nails or scalp, and a different cytokine gene expression pattern has been identified between skin and synovial tissue, explaining the differences in response to biologic therapy between these clinical areas. A predisposing genetic background, infections, obesity or biomechanical factors act as triggers and accelerate disease onset by activating macrophages, which present antigens via major histocompatibility complex type I to T cells (mainly T lymphocytes CD8) via toll-like receptor type 2. This promotes the local release of cytokines that trigger the innate and adaptive immune response.

IL-12 and TNF-α stimulate a T helper cell 1 response that releases TNF-α and INF-γ. IL-23, TNF-ß, IL-6 and IL-1b activate the T helper cell 17 response in the presence of IL-23, leading to the release of IL-17 (mainly isoform A), IL-22, IL-26 and CCL20 (macrophage inflammatory protein-3α). In addition, regulation and deactivation of the inflammatory cascade requires a T-regulatory cell mediated response via IL-2 and TNF-ß. These released cytokines interact with their transmembrane receptors, promoting the release of more cytokines and the recruitment of endothelial cells, macrophages, fibroblasts, keratinocytes, dendritic cells, epithelial cells, chondrocytes, osteoclasts and osteoblasts. Activation of the immune system results in synovitis, enthesitis, erosions and lesions of articular cartilage and skin.

Based on the literature data reviewed and the fact that Efferon CT hemoperfusion provides non-specific adsorption of excess cytokines and other inflammatory mediators, as demonstrated in numerous clinical studies,we hypothesised that cytokine sorption may have a positive clinical impact in severe and moderate forms of psoriasis. The aim of this study is to determine the efficacy and safety of anticytokine hemoperfusion using the Efferon CT device for the treatment of patients with severe and moderate psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide written informed consent and willingness and ability to comply with all requirements of the clinical trial design.
* 18 to 70 years of age.
* moderate to severe psoriasis (plaque psoriasis without psoriatic arthritis) with a disease duration of at least 6 months.
* should be receiving standard psoriasis therapy according to clinical recommendations (topical therapy, systemic therapy, phototherapy).
* Psoriasis Area and Severity Index (PASI) score ≥10,
* Body surface area (BSA) affected by psoriasis ≥10%,
* Dermatology Life Quality Index (DLQI) score >10 points,
* physician's global assessment of psoriasis severity using the static Physician Global Assessment (sPGA) ≥3 points,
* Dermatological Disease Severity Index (DIDS) score ≥2.
* for female patients: postmenopausal or have a negative pregnancy test (urinalysis) prior to enrolment. If urinalysis does not confirm absence of pregnancy, an appropriate serum analysis should be performed. The subject's pregnancy test must be negative to be eligible for inclusion in the study.

Exclusion Criteria:

* patients with other forms of psoriasis (e.g. psoriatic erythroderma, pustular psoriasis, scale psoriasis, psoriatic arthritis) or other skin conditions (e.g. eczema).
* patients on genetically engineered biological therapy (GEBT) for psoriasis.
* patients with mild forms of psoriasis.
* patients with HIV infection, syphilis, acute infectious diseases, tuberculosis.
* patients with oncological diseases.
* patients with chronic diseases in the stage of decompensation.
* patients with thrombosis and recurrent thromboembolism, thrombophlebitis.
* female patients who are pregnant or breastfeeding.
* age of patients younger than 18 years and older than 70 years.
* in the opinion of the investigator, inability of the subject to participate in this study for any other reason.
* mental condition in which the subject is unable to understand the nature, purpose and possible implications of this research.
* history of allergy, hypersensitivity to components of the extracorporeal circuit.
* inability or unwillingness to undergo all follow-up procedures until the end of the study and/or unwillingness to allow access to their medical records in accordance with national regulatory requirements at the time of consent.
* Charlson Index score greater than 6.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change in PASI (Psoriasis Area and Severity Index) score | 0 - 90 days
  Amount of PASI value reduction, %
Change in BSA (Body surface area) score | 0 - 90 days
  Amount of BSA value reduction, %
Change in the Dermatology Life Quality Index (DLQI) score | 0 - 90 days
  Amount of DLQI value reduction, %

SECONDARY OUTCOMES:
Effect of hemoperfusion using Efferon CT on the severity of pruritus according to the Visual Analogue Scale (VAS) | 0-90 days
  Change in Visual Analogue Scale (VAS) score, %
Researchers' satisfaction with treatment efficacy and side effects of Efferon CT device in treating psoriasis patients | 1-90 days
  Continuous Hemoperfusion Index-Effectiveness Index (CGI-E)
Safety of the Efferon CT device in patients with psoriasis | 1-14 days
  Frequency of incidents and adverse events
Researchers' global impression with the use of the Efferon CT device in the treatment of patients with psoriasis | 1-90 days
  Global Improvement Scale (CGI-I)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Raznatovsky, PhD, MD, Principal Investigator — North-Western State Medical University named after I.I. Mechnikov (NWSMU)
Locations (2):
- Russia (2):
  - North-Western district scientific and clinical center named after L. G. Sokolov Federal Medical and Biological Agency, Saint Petersburg
  - North-Western State Medical University named after I.I. Mechnikov (NWSMU), Saint Petersburg